CLINICAL TRIAL: NCT06577454
Title: Measuring the Effects of Neurostimulation on Risky and Ambiguous Decision-Making Capacity in People With and Without Substance Use Disorder
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Study on hold - participant recruitment suspended due to staffing limitations.
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 10001866; 001866-DA
Record Dates: First submitted 2024-08-23; First posted 2024-08-29 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-12-23

CONDITIONS: Opioid Use Disorder; Healthy Volunteers
Keywords: Opioid use Disorder; Transcranial Magnetic Stimulation (TMS); Theta Burst Stimulation (TBS); Risky decision-making
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Active TMS (Active Comparator): Participants will be blinded as to which sessions involve active TMS or sham. Those study staff involved in interacting with the participant will also be blinded. Participants will be randomized into either active-sham or sham-active session order.
  Interventions: Device: TMS (MagVenture MagPro 100 with MagOption)
- Sham TMS (Sham Comparator): Participants will be blinded as to which sessions involve active TMS or sham. Those study staff involved in interacting with the participant will also be blinded. Participants will be randomized into either active-sham or sham-active session order.
  Interventions: Device: TMS (MagVenture MagPro 100 with MagOption)

INTERVENTIONS:
Device: TMS (MagVenture MagPro 100 with MagOption) — TMS will be applied using the MagVenture MagPro 100 with MagOption (MagVenture Inc, Alpharetta, GA) stimulator with a figure-of-8 TMS coil.

SUMMARY:
Background:

The purpose of this study is to understand how a type of brain stimulation, transcranial magnetic stimulation (TMS), may help those who use opioids such as heroin or methadone. TMS uses brief magnetic pulses to affect brain activity, and is approved by the FDA to treat some mental health problems and substance use. We will evaluate how TMS may help make it easier to make certain kinds of decisions that could help one manage their opioid use. Our findings may provide support for the use of brain stimulation as a treatment to reduce opioid use.

Objective:

To understand how TMS affects brain activity associated with decision making in people who do and do not use opioids.

Eligibility:

People aged 18 to 60 years with an OUD. Healthy volunteers are also needed.

Design:

Participants will have up to 3 clinic visits over 1 to 3 months.

All participants will be screened to check if they are eligible to take part in this study. This study is completed in two parts. All eligible participants will complete the first part of the study. In the first part, you will receive one baseline magnetic resonance imaging (MRI) scan so we can take pictures of your brain while you complete computer tasks in the scanner. In these tasks, you will be asked to identify colors of words, view different images and play a game in which you can win money. If you can safely receive TMS, you will be invited to complete the second part of the study. In this part of the study, you will receive TMS and MRI over 2 sessions. For TMS, a coil will be placed on your head and a short electrical current will pass through the coil to create a magnetic pulse that stimulates your brain. You will also repeat the MRI scan and computer tasks. During one of the TMS visits you will receive active or real TMS. In the other, you will receive sham or placebo TMS, which feels like real TMS but does not affect the brain. You will receive both types of TMS. In all sessions, your urine and breath will be tested for drugs and alcohol, and you will complete questionnaires about mood and health.

DETAILED DESCRIPTION:
Study Description:

Risky decision-making is a core feature of substance use disorders and contributes to the compulsive behaviors seen in opioid use disorder (OUD). Risky decision-making can be separated into two distinct components: tolerance for known risks; and tolerance for unknown ambiguous risks. Tolerance for ambiguity in decision-making has been associated with increased risk of relapse in OUD, however conventional treatments for OUD rarely consider and target the dissociable components of decision-making that might underlie risky behaviors. In this study, we will utilize connectivity-based transcranial magnetic stimulation to selectively modulate ambiguity tolerance in decision-making in people with an OUD. Individualized cortical targets for stimulation will be derived from a baseline measurement of decision-making capacity. The ability for transcranial magnetic stimulation (TMS) to modulate ambiguity tolerance in decision-making will be assessed (relative to placebo stimulation), as well as clinical correlates, such as craving.

Objectives:

* Primary Objectives:

  * Determine neural correlates of risk and ambiguity tolerance in healthy controls and people with OUD.
  * Measure the impact of a type of TMS (theta burst stimulation) on ambiguity tolerance in healthy controls and people with OUD.
* Secondary Objectives:

  * Determine the impact of TMS on resting-state brain activity.
  * Determine the impact TMS on outcomes that are relevant to substance use and relapse (e.g., craving).
* Tertiary/Exploratory Objectives:

  * The effect of sex on the above metrics will be explored.

Endpoints:

The impact of transcranial magnetic stimulation on decision making will be assessed several ways.

* Primary Endpoints:

  * Brain reactivity during decision-making task that separates tolerance for risk and tolerance for ambiguity.
  * Modulation of behavior and neural activity in areas of the brain associated with ambiguity tolerance by TMS.
* Secondary Endpoints:

  * The influence of TMS on the brain s resting state function will be assessed.
  * The influence of TMS on substance use-related outcomes will be assessed.
* Tertiary/Exploratory Endpoints:

  * Completion of baseline visit where neuromodulation is not administered.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

Both groups:

-Participants will be volunteers between the ages of 18-60.

Opioid-using group:

* Participants must meet DSM-5 criteria for an opioid use disorder (active or in remission and on maintenance therapy).
* Participants must be currently enrolled in and receiving medication-assisted treatment for opioid use disorder (MOUD; such as methadone, buprenorphine or naltrexone) and report a stable dose of their medication for at least 4 weeks prior to enrollment.*
* Participants in this group can meet DSM-5 criteria for other substance use disorders (such as alcohol, nicotine, or cocaine use disorder) currently or in the past but must also meet criteria for an OUD.

  * To note, participants in the opioid-using group will not receive direct clinical care from NIDA study staff, but enrollment in a MOUD program will be required for inclusion in this study. This will be assessed by self-report of enrollment in a known MOUD program and a urine screen confirming their reported treatment. Participants will also sign a release of information (ROI) form that provides contact details for their treatment provider and allows for communication between the study team and the participants treatment provider if necessary.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

Controls:

-Participants cannot meet DSM-5 criteria for current substance use disorders other than nicotine and marijuana and cannot meet criteria for current moderate or severe alcohol use disorder.

All participants:

* Participants cannot meet DSM-5 criteria for lifetime and/or current psychotic disorders such as bipolar disorder, schizophrenia, schizoaffective disorder.
* Participants cannot have a history of major head trauma resulting in cognitive impairment, seizure, or other neurological disorders.
* Participants cannot have any history of significant neurological disorders, including seizures, epilepsy, or cognitive impairment which may impact MRI metrics. MAI will use discretion in evaluating the impact of minor events or history reported.
* Participants cannot be pregnant.
* Participants with Major Depressive Disorder (per DSM-V criteria) must be stable on medication(s) for 3 months.
* Subjects with suicidal ideation where outpatient treatment is determined unsafe.
* Subjects that cannot speak English. Justification: To include non-English speakers, we would have to translate the consent and other study documents and hire and train bilingual staff, which would require resources that we do not have and could not justify, given the small sample size for each experiment. Additionally, the data integrity of some of the cognitive tasks and standardized questionnaires used in this study would be compromised as they have only been validated in English. Most importantly, ongoing communication regarding safety procedures is necessary when participants are undergoing MRI procedures. The inability to effectively communicate MRI safety procedures in a language other than English could compromise the safety of non-English speaking participants.
* Any contraindications to MRI.
* For subjects continuing to the TMS portion of the protocol, contraindications for TMS.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2027-08-06 (Estimated); Study Completion 2027-08-06 (Estimated)

PRIMARY OUTCOMES:
Determine neural correlates of risk and ambiguity tolerance in healthy controls and people with OUD. | 1-3 months
  Preliminary works demonstrates that neural correlates of risk and ambiguity tolerance are separable
Measure the impact of transcranial magnetic stimulation (TMS) on ambiguity tolerance in healthy controls and people with OUD | 1-3 months
  TMS has been used to modulate brain activity in areas associated with decision-making

SECONDARY OUTCOMES:
Determine the impact of TMS on resting-state brain activity | 1-3 months
  There is evidence that resting state brain organization/function influences task activation. Whether TMS impacts resting state networks associated will be tested.
Determine the impact TMS on outcomes that are relevant to substance use and relapse (e.g., craving) | 1-3 months
  TMS has been shown to modulate clinical endpoints associated with drug use. The influence of TMS on craving will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Amy C Janes, Ph.D., Principal Investigator — National Institute on Drug Abuse (NIDA)
Locations (1):
- National Institute on Drug Abuse, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Some information collected under this protocol may be placed into one or more scientific databases after it has been stripped of identifiers such as name, so that it may be used for future research on any topic and shared broadly for research purposes. A researcher who wants to study the information must apply to the database and be approved. Researchers with an approved study may be able to see and use the data from this protocol, along with that from many other studies. We do not expect any direct benefits for participants resulting from the use of protocol data and information, though new discoveries that may help other people could occur. The Principal Investigator is open to answering any participant questions about how these data may be used.